CLINICAL TRIAL: NCT05380531
Title: Personalized Perioperative Analgesia Platform (PPAP) for Cesarean Section
Acronym: PPAP C-Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Senthil Sadhasivam (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Senthil Sadhasivam, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21100167; 1U01TR003719-01A1 (NIH)
Record Dates: First submitted 2022-04-19; First posted 2022-05-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section Complications; Opioid Use
Keywords: Opioid Exposure

STUDY DESIGN:
Intervention Model Description: Interventional study with mother undergoing elective c-section and the infant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mother undergoing planned Cesarean section (Experimental): Mother subject will have genotyping blood draw performed at the time of controlled delivery (CD). Blood samples and breast milk samples will also be taken during the oxycodone dosing schedule.
  Interventions: Diagnostic Test: Preoperative Genotyping
- Infant (Experimental): Infant subject will have genotyping blood draw performed only at the time of controlled delivery (CD)
  Interventions: Diagnostic Test: Preoperative Genotyping

INTERVENTIONS:
Diagnostic Test: Preoperative Genotyping — Genotype based risk prediction and personalized pain management

SUMMARY:
The purpose of this collaborative CTSA (Clinical and Translational Science Award) application is to develop an innovative perioperative precision analgesia platform (PPAP) to improve analgesia and reduce serious immediate and long-term adverse outcomes of perioperative opioids in breastfeeding mothers and their infants

DETAILED DESCRIPTION:
The approach includes 1) development and implementation of an innovative PPAP infrastructure at participating CTSA hubs (Aim 1) and 2) to improve analgesia and reduce serious immediate and long-term adverse outcomes of perioperative opioids and precision dosing in nursing mothers and infants (Aim 2).

SPECIFIC AIMS: The purpose of this collaborative CTSA application is to develop an innovative perioperative precision analgesia platform (PPAP) to improve analgesia and reduce serious immediate and long-term adverse outcomes of perioperative opioids in

Aim 1. Develop and implement a perioperative precision analgesia platform (PPAP) by linking genomics to opioid metabolism, Clinical Pharmacogenetics Implementation (CPIC) guidelines, precision dosing, clinical safety, and personalizing analgesia

Aim 2. Evaluate utility of PPAP in nursing mothers and their newborns following Cesarean Section The investigators hypothesize that CYP2D6 and other (ABCB1, and OPRM1) variants will explain clinical and pharmacokinetic variations of oxycodone, and PPAP implementation will reduce adverse effects in mothers and infants.

ELIGIBILITY:
Inclusion Criteria:

Adult women (>18 yr) All races American Society of Anesthesiologists Classification (ASA) physical status: 1 to 3 undergoing elective Cesarean section that are willing to receive in-patient opioids.

Exclusion Criteria:

1. Health conditions including uncontrolled diabetes (gestational or pre-existing) or hypertension (pre-eclampsia, eclampsia, or chronic)
2. Any history of opioid misuse before or during pregnancy-per self-report and clinical notes
3. Preoperative severe pain and opioid use/misuse, allergy to oxycodone
4. Allergy to oxycodone
5. Significant neurological disorders, liver and renal diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Look at genetic factors predisposing patients to immediate postoperative opioid-adverse effects Respiratory Depression (RD) and Postoperative Nausea and Vomiting (PONV) | Immediately post-surgery during hospital stay
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with patients who experience RD and PONV in the immediate post-surgical period (4 days) in the hospital
Look at genetic factors predisposing patients to immediate postoperative opioid-adverse effects Respiratory Depression (RD) and Postoperative Nausea and Vomiting (PONV) | At home up to 1 year post-surgery
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with patients who experience RD and PONV in the post-surgical period at home up to 1-year
Look at genetic factors predisposing patients to inadequate surgical pain relief with oxycodone | Immediately post-surgery during hospital stay
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with patients who experience poor pain relief in the immediate post-surgical period (4 days) in the hospital. Poor pain relief will be measured using the Numerical Rating Scale (NRS), which runs on a 0-10 scale; 0 being no pain at all, 10 being the worst pain imaginable.
Look at genetic factors predisposing patients to inadequate surgical pain relief with oxycodone | At home up to 1 year post-surgery
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with patients who experience poor pain relief in the post-surgical period at home up to 1-year. Poor pain relief will be measured using the Numerical Rating Scale (NRS), which runs on a 0-10 scale; 0 being no pain at all, 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Look at the impact of CYP2D6 variants on oxycodone's clinical dosing in patients to see if specific variants correlate with a need for lower or higher doses of analgesic. | Pre-operative to post-operative day 2
  The investigators will look at CYP2D6 variants to find correlations in oxycodone's PK sampling and the need for dose adjustments that lead to desired clinical outcomes in women undergoing a cesarean section and their infant.

OTHER OUTCOMES:
Look at OPRM1 epigenetics and OPRM1, FAAH, GCH1, DRD2 variants to find correlations with chronic persistent surgical pain (CPSP) up to 1-year post-surgery | Post-operative up to 1-year
  Patients will be asked to complete psychological questionnaires post-surgery to assess psycho-psychological factors that may correlate with CPSP. CPSP is defined as pain that develops after a surgical procedure and lasts at least 3 months and significantly affects health-related quality of life.
Look at OPRM1 epigenetics and OPRM1, FAAH, GCH1, DRD2 variants to find correlations with opioid dependence (OD) up to 1-year post-surgery | Post-operative up to 1-year
  Patients will be asked to complete psychological questionnaires post-surgery to assess psycho-psychological factors that may correlate with opioid dependence (OD). OD will be determined using the validated Sophia Observation Withdrawal Symptoms Scale (SOS). The SOS is based on a 15-point scale.
Look at OPRM1 epigenetics and OPRM1, FAAH, GCH1, DRD2 variants to find correlations with opioid dependence (OD) up to 1-year post-surgery | Post-operative up to 1-year
  Patients will be asked to complete psychological questionnaires post-surgery to assess psycho-psychological factors that may correlate with opioid dependence (OD). OD will be determined using the Clinical Opiate Withdrawal Scale (COWS). The COWS is based on a scale with a minimum score of 5 and maximum score of 48; 5-12 = mild, 13-24 = moderate, 25-36 = moderately severe, more than 36 = severe withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Sadhasivam, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Magee Women's Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No current IPD sharing plan anticipated